CLINICAL TRIAL: NCT03214640
Title: Evaluation of Success in Neuraxial Block Placement Between Using Palpation of Landmark Versus Pocket-Size Handheld Ultrasound (U/S) Method
Brief Title: Rivanna Ultrasound for Neuraxial Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00044968
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-03

CONDITIONS: Analgesia
Keywords: neuraxial analgesia; spinal block; epidural block
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: There are 4 arms for this study--two are active comparators and two are experimental. The first arm is palpation with spinal block. The second arm is palpation with neuraxial block. The third arm is ultrasound with spinal block. The fourth arm is ultrasound with neuraxial block. Randomization is done twice - first for randomization of spinal block subjects between using palpation versus ultrasound method; and again randomization for neuraxial block (combined spinal epidural) subjects between using palpation versus ultrasound method. There will be a total of 120 planned evaluable subjects. This consists of planned evaluable randomized 60 subjects receiving spinal block for cesarean delivery (30 for palpation and 30 for ultrasound); and planned evaluable randomized 60 subjects receiving neuraxial (combined spinal epidural) block for labor analgesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Palpation with spinal block (Group C-P) (Active Comparator): insertion will be identified by palpation using conventional landmarks (spinous process and iliac crest) for placement of spinal block for cesarean delivery
  Interventions: Other: Palpation; Procedure: Spinal Block
- Palpation with neuraxial block (Group L-P) (Active Comparator): the needle insertion site for the neuraxial block will be identified with palpation for labor analgesia, using the spinous process and iliac crest for reference
  Interventions: Other: Palpation; Procedure: Neuraxial Analgesia
- Rivanna Accuro Ultrasound Device with spinal block (Group C-R) (Experimental): insertion will be identified with Rivanna Accuro U/S device for placement of spinal block for cesarean delivery
  Interventions: Device: Rivanna Accuro US Device; Procedure: Spinal Block
- Rivanna Ultrasound Device with neuraxial block (Group L-R) (Experimental): insertion will be identified with Rivanna Accuro U/S device for placement of neuraxial block (combined spinal epidural) for labor analgesia
  Interventions: Device: Rivanna Accuro US Device; Procedure: Neuraxial Analgesia

INTERVENTIONS:
Device: Rivanna Accuro US Device — When the subject is ready for neuraxial procedure, the location for the epidural or spinal needle insertion will be identified with Rivanna Accuro U/S device. For subjects in group C-R or L-R, the needle insertion site will be the site identified by the Rivanna Accuro U/S device. After placement of spinal for Cesarean or epidural for labor, the usual standard dose of medication will be administered as in usual manner for patients regardless in this study or not.
  Arms: Rivanna Accuro Ultrasound Device with spinal block (Group C-R); Rivanna Ultrasound Device with neuraxial block (Group L-R)
Other: Palpation — When the subject is ready for neuraxial procedure, the location for the epidural or spinal needle insertion will be identified with Palpation method using conventional landmarks (spinous process and iliac crest). For subjects in group C-P or L-P, the needle insertion site will be the site identified by the Palpation method. After placement of spinal for Cesarean or epidural for labor, the usual standard dose of medication will be administered as in usual manner for patients regardless in this study or not.
  Arms: Palpation with neuraxial block (Group L-P); Palpation with spinal block (Group C-P)
Procedure: Neuraxial Analgesia — Labor analgesia will be provided utilizing the standard medications to provide labor analgesia
  Arms: Palpation with neuraxial block (Group L-P); Rivanna Ultrasound Device with neuraxial block (Group L-R)
Procedure: Spinal Block — Spinal anesthetic medications will be utilized in providing surgical block for cesarean delivery as is standard of care
  Arms: Palpation with spinal block (Group C-P); Rivanna Accuro Ultrasound Device with spinal block (Group C-R)

SUMMARY:
We hypothesize that the Rivanna Accuro or similar U/S device would reduce time to success of identifying epidural and/or intrathecal spaces as compared to conventional palpation method.

DETAILED DESCRIPTION:
Administration of (neuraxial blocks) spinal and epidural blocks is commonly achieved by first palpating the landmarks for midline with spinous process and iliac crest for L3-4-5 intervertebral spaces. With an epidural block, a loss of resistance in a pressurized syringe is used to incrementally advance the epidural needle until identification of epidural space with loss of resistance in the pressurized syringe. With a spinal block, the spinal needle is advanced incrementally until a noted "feel" of dural puncture together with return of spinal fluid via the spinal needle. The palpation technique and somewhat "blind" technique to identify the spinal and epidural spaces become more difficult and less reliable particularly with the increasing prevalence of the morbid and super-morbid obese patients. Ultrasound devices have become common and successful with non-neuraxial blocks and venous accesses, both involving mostly non-bony, soft tissues. Application of conventional ultrasound for neuraxial blocks has been limited by its bulkiness, limited imaging for bony structures and lack of automated artificial intelligent algorithm for pattern recognition. Recent technological advancement has addressed the aforementioned limitations. Rivanna Accuro is one such device that has gained FDA approval and may have helped in addressing some of these issues. It is a handheld (pocket size) U/S device with real time pattern recognition for bony structures such as the spine while providing 3-D overlay for recognition of the midline spinous process and epidural spaces and distance. The investigators hypothesize that the Rivanna Accuro or similar U/S device would reduce time to success of identifying epidural and/or intrathecal spaces as compared to conventional palpation method. We will compare placement of neuraxial block between palpation method versus ultrasound method. We will compare placement of spinal block for cesarean delivery with palpation versus with ultrasound method, and then comparing placement of neuraxial analgeisa block (combined spinal epidural analgesia) for labor analgesia with palpation versus ultrasound method.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30
* Female requesting analgesia for delivery, be it via vaginal or cesarean delivery

Exclusion Criteria:

* Allergy to ultrasound gel
* Contraindication to receiving neuraxial analgesia
* Under the age of 18

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pan, MD, MSEE, Principal Investigator — Professor, Anesthesiology
Locations (1):
- Novant Health Forsyth Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: 510(k) clearance for the Rivanna Accuro handheld ultrasound device — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K132736

RESULTS

PARTICIPANT FLOW:
Groups:
- Palpation With Spinal Block (Group C-P): insertion will be identified by palpation using conventional landmarks (spinous process and iliac crest) for placement of spinal block for cesarean delivery
  Palpation description:: When the subject is ready for neuraxial procedure, the location for the epidural or spinal needle insertion will be identified with Palpation method. For subjects in group C-P or L-P, the needle insertion site will be the site identified by the Palpation method. After placement of spinal for Cesarean or epidural for labor, the usual standard dose of medication will be administered as in usual manner for patients regardless in this study or not.When the subject is ready for neuraxial procedure, the location for the epidural or spinal needle insertion will be identified by palpation using conventional landmarks (spinous process and iliac crest). Those in group P, the neuraxial block will be performed as in the usual method using the needle insertion site identified with palpation. After placement of neuraxial labor analgesia the usual standard dose of medication will be administered as in usual manner for patients regardless in this study or not.
  Spinal Block: Spinal anesthetic medications will be utilized in providing surgical block for cesarean delivery as is standard of care
- Palpation With Neuraxial Block (Group L-P): the needle insertion site for the neuraxial block will be identified with palpation for labor analgesia
  Palpation description:: When the subject is ready for neuraxial procedure, the location for the epidural or spinal needle insertion will be identified with Palpation method. For subjects in group C-P or L-P, the needle insertion site will be the site identified by the Palpation method. After placement of spinal for Cesarean or epidural for labor, the usual standard dose of medication will be administered as in usual manner for patients regardless in this study or not.When the subject is ready for neuraxial procedure, the location for the epidural or spinal needle insertion will be identified by palpation using conventional landmarks (spinous process and iliac crest). Those in group P, the neuraxial block will be performed as in the usual method using the needle insertion site identified with palpation. After placement of neuraxial labor analgesia the usual standard dose of medication will be administered as in usual manner for patients regardless in this study or not.
  Neuraxial Analgesia: Labor analgesia will be provided utilizing the standard medications to provide labor analgesia
Period: Overall Study
Arm/Group | Palpation With Spinal Block (Group C-P) | Palpation With Neuraxial Block (Group L-P) | Rivanna Accuro Ultrasound Device With Spinal Block (Group C-R) | Rivanna Ultrasound Device With Neuraxial Block (Group L-R)
Started | 31 | 32 | 31 | 34
Completed | 30 | 30 | 30 | 30
Not Completed | 1 | 2 | 1 | 4
Not completed — Protocol Violation | 1 | 2 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palpation With Spinal Block (Group C-P) | Palpation With Neuraxial Block (Group L-P) | Rivanna Accuro Ultrasound Device With Spinal Block (Group C-R) | Rivanna Ultrasound Device With Neuraxial Block (Group L-R) | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5.8) | 27.3 (5.3) | 29.8 (4.8) | 28.6 (6.4) | 29.53 (5.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female Subjects | 30 | 30 | 30 | 30 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 8 | 7 | 5 | 4 | 24
  White | 20 | 22 | 24 | 26 | 92
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 30 | 120

OUTCOME MEASURES:

1. Primary Outcome: Time to Success of Neuraxial Block Placement
Description: Time it takes to successfully identify the epidural space (defined by loss of resistance) for the groups of subjects receiving labor neuraxial analgesia; and spinal fluid flow into the hub of spinal needle for the groups of subjects receiving cesarean spinal anesthetic - length of time (in minutes) it takes to get block placed, between palpation and ultrasound groups among patients with labor neuraxial analgesia patients and cesarean spinal anesthetic, respectively and spinal fluid flow with spinal needle - length of time (in seconds) it takes to get block placed, between the 2 groups.
Time Frame: 60-225 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Palpation With Spinal Block (Group C-P) | Palpation With Neuraxial Block (Group L-P) | Rivanna Accuro Ultrasound Device With Spinal Block (Group C-R) | Rivanna Ultrasound Device With Neuraxial Block (Group L-R)
Number analyzed (Participants) | 30 | 30 | 30 | 30
seconds | 122 [60 to 225] | 111 [72.7 to 211] | 50 [26 to 106] | 78.5 [48.7 to 115.5]

2. Secondary Outcome: Total Number of Needle Passes Per Placement
Description: Number of needle Passes before successful placement
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: number of needle passes needed to succes
Arm/Group | Palpation With Spinal Block (Group C-P) | Palpation With Neuraxial Block (Group L-P) | Rivanna Accuro Ultrasound Device With Spinal Block (Group C-R) | Rivanna Ultrasound Device With Neuraxial Block (Group L-R)
Number analyzed (Participants) | 30 | 30 | 30 | 30
number of needle passes needed to succes | 2 [1 to 4] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 1]

3. Secondary Outcome: Needle Passing Success at First Attempt
Description: Number of times of success (Number of patients) with first (single) attempt needle pass success
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Palpation With Spinal Block (Group C-P) | Palpation With Neuraxial Block (Group L-P) | Rivanna Accuro Ultrasound Device With Spinal Block (Group C-R) | Rivanna Ultrasound Device With Neuraxial Block (Group L-R)
Number analyzed (Participants) | 30 | 30 | 30 | 30
participants | 10 | 18 | 18 | 24

ADVERSE EVENTS:
Time Frame: Time frame of monitoring AEs and SAEs was from time of enrollment to 24 hours post delivery
Description: Study staff looked for postdural puncture headaches, neurological injury, or other serious events such as significant cv pul neurological and systemic complications. Study staff followed all Subjects the next day within 24 hours after delivery to make sure no untoward event no AR or SAEs.
Arm/Group | Palpation With Spinal Block (Group C-P) | Palpation With Neuraxial Block (Group L-P) | Rivanna Accuro Ultrasound Device With Spinal Block (Group C-R) | Rivanna Ultrasound Device With Neuraxial Block (Group L-R)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT03214640/Prot_SAP_001.pdf
  • Informed Consent Form (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03214640/ICF_000.pdf